CLINICAL TRIAL: NCT06175416
Title: Spontaneous Pneumothorax in Adolescents: Inventory and Management
Brief Title: Spontaneous Pneumothorax in Adolescents
Acronym: PNSA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8700
Record Dates: First submitted 2022-09-13; First posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Pneumothorax, Spontaneous
Keywords: Pneumothorax; Spontaneous; Pleural cavity
MeSH Terms: conditions — Pneumothorax

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pneumothorax is characterized by an abnormal presence of air in the pleural cavity, that is to say between the two layers of the pleura, the membrane that surrounds the lungs and lines the rib cage. "The patient is usually seized with sudden chest pain and difficulty in breathing.

In this retrospective research, the investigators wish to carry out an inventory of the management of spontaneous pneumothorax in adolescents within the University Hospitals of Strasbourg

ELIGIBILITY:
Inclusion criteria:

* Adult patient (18-20 years old)
* Minor patient aged 14-17 years old
* Any gender
* Spontaneous pneumothorax without apparent cause, between 14 and 20 years old
* Patient operated on at the HUS between 2010 and 2021
* Patient not objecting to the reuse of their data for scientific research purposes.
* Holders of parental authority who do not object to the reuse of their child's data for scientific research purposes.

Exclusion criteria:

* Patient who has expressed his opposition to the reuse of his data for scientific research purposes.
* Holders of parental authority who have expressed their opposition to the reuse of their child's data for scientific research purposes.
* Secondary origin of the pathology: Cystic fibrosis, postoperative pneumothorax, post-traumatic,
* Subject having been treated initially in another structure without further information.

Ages: 14 Years to 20 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patient (aged between 14-20 years old) having pontaneous pneumothorax without apparent cause and operated on at the HUS between 2010 and 2021.
Sampling Method: Non-Probability Sample
Enrollment: 134 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Retrospective description of the management of spontaneous pneumothorax in adolescents in the Strasbourg University Hospital | Files analysed retrospectively from January 1, 2010 and December 31, 2021 will be examined
  This study is retrospective, the analysis focuses on the medical records of patients treated at the Strasbourg University Hospital between between January 1, 2010 and December 31, 2021.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Chirurgie pédiatrique - CHU de Strasbourg - France, Strasbourg, France